CLINICAL TRIAL: NCT06811831
Title: Evaluation of the Efficacy of MACitentan in the Treatment of CoronaryMICrovascular Angina: a Pilot Study
Brief Title: Evaluation of the Efficacy of MACitentan in the Treatment of CoronaryMICrovascular Angina (MACMIC)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingang Zheng, Head of Department of Cardiology, China-Japan Friendship Hospital, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-KY-0501
Record Dates: First submitted 2025-01-22; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Coronary Microvascular Angina; Macitentan
Keywords: coronary microvascular angina; angina with non-obstructive coronary arteries; Macitentan; Endothelin-receptor antagonists
MeSH Terms: interventions — macitentan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Taking Macitentan Group (Experimental)
  Interventions: Drug: Macitentan 10 mg tablet, once daily.

INTERVENTIONS:
Drug: Macitentan 10 mg tablet, once daily. — After the patient signed an informed consent form, Macitentan was given as an oral medication (10 mg once daily) for a period of 4 weeks

SUMMARY:
Coronary microvascular angina (MVA) significantly reduces quality of life and increases the risk of heart problems in patients with angina. Unfortunately, there are no effective treatments available yet. The endothelin-1 (ET-1) - endothelin receptor (ETRs) system plays a critical role in MVA. Preclinical studies demonstrate that ETRs antagonists or pericyte-specific knockdown of ETRs can improve coronary microvascular function in myocardial ischemia/reperfusion mice and diabetic mice. Foreign clinical drug trials have shown that ETRs antagonists may alleviate patients' symptoms. However, these studies predominantly rely on conventional coronary angiography rather than direct assessment of coronary microvascular function. Early experimental trials using ETRs antagonists reported a high incidence of side effects, such as sodium retention and headaches, which negatively impacted treatment satisfaction.

To address these limitations, a pilot study is proposed to evaluate the efficacy of macitentan in MVA treatment. This investigation will implement thermodilution-based coronary microcirculation function testing to precisely characterize the severity and subtype of coronary microvascular lesions in MVA patients. By administering macitentan - a safer ETRs antagonist - the study aims to systematically assess improvements in coronary microvascular function, angina symptom relief, and adverse event incidence. The findings are expected to provide critical evidence regarding the therapeutic potential and safety profile of macitentan, while establishing foundational data for subsequent large-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old.
* With typical angina symptoms.
* Excluding obstructive coronary lesions (coronary stenosis ≤50% or FFR ≥0.8) by CAG.
* Coronary microcirculatory function CFR<2.5 and/or IMR>25 assessed by temperature dilution method.

Exclusion Criteria:

* Pregnant or lactating women.
* History of heart attack within the last 90 days.
* Severe heart disease (e.g., moderate to severe heart failure, severe heart valve disease).
* Severe renal impairment (GFR <30 ml/min/1.73m2).
* Severe liver disease (Child-Pugh class C).
* Moderately severe anaemia (haemoglobin concentration <90 g/L).
* Participation in another drug intervention trial study within the last 90 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Week 4 in the Coronary Microcirculatory Function Indices Assessed by CFR and IMR | the duration of hospital stay, an expected average of 2 weeks; 4-week follow-up
  Coronary microcirculatory function indices include Coronary Flow Reserve (CFR) and Index of Microcirculatory Resistance (IMR)
  1. Coronary Flow Reserve (CFR): A unitless ratio quantifying maximal coronary blood flow augmentation capacity, measured via thermodilution as the ratio of hyperemic to resting coronary flow. The commonly used cut-off value is 2.0 or 2.5. Increased ratio indicates improved microvascular dilation capacity
  2. Index of Microcirculatory Resistance (IMR): A pressure-derived metric (units: mmHg·s) assessing microvascular resistance using thermodilution, calculated as distal coronary pressure multiplied by mean transit time during maximal hyperemia. The commonly used cut-off value is 25. Decreased value indicates reduced microvascular resistance

SECONDARY OUTCOMES:
Change in Score of the Seattle Angina Questionnaire (SAQ) | the duration of hospital stay, an expected average of 2 weeks; 4-week follow-up; 8-week follow-up
  The Seattle Angina Questionnaire (SAQ) is a 19-item instrument designed to assess the impact of angina on patients' daily lives across five domains: physical limitation, angina stability, angina frequency, treatment satisfaction, and disease perception. Each item is scored on a 0-100 scale, where higher scores indicate fewer symptoms and better quality of life.
Change in Angina Symptoms Assessed by Angina Diary | the duration of hospital stay, an expected average of 2 weeks; 4-week follow-up; 8-week follow-up
  The angina diary is a structured log where patients record angina episodes, including their frequency, severity, duration, and possible triggers. Symptom severity is classified using a 4-level grading system similar to the Canadian Cardiovascular Society (CCS) angina.
Change in the Score of 6-minute Walking Distance (6MWD) | the duration of hospital stay, an expected average of 2 weeks; 4-week follow-up; 8-week follow-up
  The 6MWD test evaluates functional exercise capacity by measuring the total distance a patient can walk on a flat surface in 6 minutes. The test reflects cardiovascular fitness and symptom severity.
Incidence of rehospitalisation for angina or heart failure. | 4-week follow-up; 8-week follow-up

OTHER OUTCOMES:
Safety Outcome | 8-week follow-up
  Occurrence of all adverse events such as hydrosodium storage, anaemia, headache and hypotension et al.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China